CLINICAL TRIAL: NCT05354258
Title: Feasibility and Effectiveness of Delivering Mass Drug Administration for Helminths Through the Seasonal Malaria Chemoprevention (SMC) Platform in a West African Paediatric Population
Brief Title: Feasibility and Safety of Combining Anti-malarial With Deworming Drugs in African Children
Acronym: MALHELMIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Université de Thies, UFR Santé, Senegal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26770
Record Dates: First submitted 2022-04-12; First posted 2022-04-29 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-04

CONDITIONS: Malaria; Soil Transmitted Helminths; Schistosomiasis; Integrated Control; Seasonal Malaria Chemoprevention; Mass Drug Administration With Anthelminthic Drugs
MeSH Terms: conditions — Malaria; Schistosomiasis | interventions — Albendazole; Praziquantel; Amodiaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin A + Zinc supplements on Day 0, followed by SMC course on Day 1,2 & 3 (Placebo Comparator)
  Interventions: Drug: Amodiaquine; Drug: Sulfadoxine pyrimethamine
- Praziquantel + Vitamin A on Day 0, followed SMC course on Days 1,2 & 3 (Experimental)
  Interventions: Drug: Praziquantel; Drug: Amodiaquine; Drug: Sulfadoxine pyrimethamine
- Albendazole + Praziquantel on Day 0, followed by SMC course on Days 1, 2 & 3 (Experimental)
  Interventions: Drug: Albendazole; Drug: Praziquantel; Drug: Amodiaquine; Drug: Sulfadoxine pyrimethamine

INTERVENTIONS:
Drug: Albendazole — Anthelminthic drugs for the treatment of soil-transmitted helminths
  Arms: Albendazole + Praziquantel on Day 0, followed by SMC course on Days 1, 2 & 3
Drug: Praziquantel — Anthelminthic drugs for the treatment of schistosomiasis
  Arms: Albendazole + Praziquantel on Day 0, followed by SMC course on Days 1, 2 & 3; Praziquantel + Vitamin A on Day 0, followed SMC course on Days 1,2 & 3
Drug: Amodiaquine — SMC partner drug
Drug: Sulfadoxine pyrimethamine — SMC partner drug

SUMMARY:
Malaria remains a major health problem, especially in sub-Saharan Africa where more than 90% of the disease and deaths occur in children. Adding to this high burden among the children is the co-existence of intestinal and genito-urinary worms. Prominent among these are soil-transmitted helminths and schistosomiasis. Existing control programmes for the worms are operating below the expected level, despite the commitments and support that followed the 2012 London Declaration of achieving 75% treatment coverage by 2020. On the other hand, a malaria prevention programme, called Seasonal Malaria Chemoprevention (SMC), introduced in the same year 2012 has achieved more than 75% treatment coverage and prevented 75-85% cases of uncomplicated and severe malaria in children. This encouraging development supports the need to explore the strategies involving the integration of worm control with successful platforms such as SMC. This would align worm and malaria control with the WHO road map for Neglected Tropical Diseases (NTD) of ending the neglect to attain Sustainable Development Goals by eradicating diseases of poverty and promoting health and well-being for those at risk. Given this context, it is important to develop a treatment approach that combines malaria and helminth control in an integrated framework that will be safe, effective and easy to deliver. This study will, therefore, investigate the feasibility and effectiveness of co-administration of anthelminthic and SMC drugs in a high-risk paediatric population living in a malaria-helminth co-endemic setting in Senegal, West Africa. This study is designed to test the hypothesis that co-administration of SMC and anthelminthic drugs will be safe and tolerated among children aged 1-14 years and that the incidence of side effects will not be significant. The objectives of this study are to assess the safety, tolerability, and effects of co-administration of SMC and anthelminthic drugs among the children

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 1-14 years;
* Provision of a written informed consent by the parent/caregiver and a positive assent by children aged ≥ 12 years (in line with legal regulations in Senegal);
* Willingness to provide finger-prick blood samples, urine, and stool samples;
* Residence in the study area for at least six months

Exclusion Criteria:

* Acutely ill child at the time of the drug administration;
* Child whose parents/caregivers decline to provide consent;
* A known HIV positive child receiving cotrimoxazole prophylaxis;
* A child who has received a dose of any of sulphadoxine-pyrimethamine, amodiaquine, albendazole or praziquantel during the previous six months;
* A child with a known allergy to any of sulphadoxine-pyrimethamine, amodiaquine, albendazole or praziquantel.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | For six consecutive days after start of the drug administration
  Incidence of Treatment-Emergent Adverse Events will be measured by collecting solicited and unsolicited adverse events and adverse drug reactions for causal relationships to the study drugs.

SECONDARY OUTCOMES:
Prevalence of helminth co-infection | On the day of randomisation (pre-intervention) and up to 4 months post-intervention
  Faecal egg counts for soil transmitted helminths
Prevalence of Schistosoma co-infection | On the day of randomisation (pre-intervention) and up to 4 months post-intervention
  Urine egg counts for Schistosoma haematobium
Prevalence of intensity of helminth infection | On the day of randomisation (pre-intervention) and up to 4 months post-intervention
  Arithmetic mean intensity of helminth infection

OTHER OUTCOMES:
Prevalence of anaemia | On the day of randomisation (pre-intervention) and up to 4 months post-intervention
  Haemoglobin concentration of all study children will be checked using HemoCue®

CONTACTS AND LOCATIONS:
Overall Officials: Brian Greenwood, MD, FMedSci, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Saraya Health Centre, Saraya, Région de Kédougou, Senegal

IPD SHARING:
Plan to Share IPD: Yes
We will share the summary results of this trial or a link to the summary results within the trial registration record within 12 months of the study completion date
Supporting Information: Study Protocol
Time Frame: Within 12 months of the study completion date
Access Criteria: Open access requests will be entertained, the decision will be made by the Principal Investigator, quality of the request will be reviewed before granting it

REFERENCES:
- [Derived] Afolabi MO, Sow D, Agbla SC, Fall EHB, Sall FB, Seck A, Manga IA, Mbaye IM, Loum MA, Camara B, Niang D, Gueye B, Sene D, Kane NM, Diop B, Diouf A, Gaye NA, Diouf MP, Lo AC, Greenwood B, Ndiaye JLA. Feasibility and safety of integrating mass drug administration for helminth control with seasonal malaria chemoprevention among Senegalese children: a randomized controlled, observer-blind trial. Malar J. 2023 Nov 13;22(1):348. doi: 10.1186/s12936-023-04784-z. PMID 37957702
- [Derived] Afolabi MO, Diaw A, Fall EHB, Sall FB, Diedhiou A, Seck A, Camara B, Niang D, Manga IA, Mbaye I, Sougou NM, Sow D, Greenwood B, Ndiaye JLA. Provider and User Acceptability of Integrated Treatment for the Control of Malaria and Helminths in Saraya, South-Eastern Senegal. Am J Trop Med Hyg. 2023 Sep 18;109(5):1047-1056. doi: 10.4269/ajtmh.23-0113. Print 2023 Nov 1. PMID 37722662
- [Derived] Afolabi MO, Sow D, Ndiaye JLA, Greenwood B. Safety and effectiveness of delivering mass drug administration for helminths through the seasonal malaria chemoprevention platform among Senegalese children: study protocol for a randomised controlled trial. Trials. 2022 Aug 3;23(1):627. doi: 10.1186/s13063-022-06579-0. PMID 35922819